CLINICAL TRIAL: NCT00578721
Title: Phase IIA Clinical Biomarker Trial of Aspirin and Arginine Restriction in Colorectal Cancer Patients
Brief Title: Trial of Aspirin and Arginine Restriction in Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jason Zell, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UCI 07-47 HS# 2007-5892
Record Dates: First submitted 2007-12-18; First posted 2007-12-21 (Estimated); Results first posted 2023-06-26 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; aspirin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 325 mg Aspirin (Experimental): 325 mg aspirin po qd with arginine-restricted diet
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 325 mg taken daily with an arginine-restricted diet

SUMMARY:
The purpose of this research study is to understand the effects of oral aspirin taken daily with an arginine-restricted diet on certain colorectal cancer biomarkers in treated colorectal cancer patients. Patients with colorectal cancer are at high risk for recurrence and for development of secondary colorectal cancers in the future. Specific chemicals (polyamines, prostaglandins) in the body referred to as biomarkers can be measured to help understand a person's risk for developing colorectal cancer. Specific biomarkers associated with colorectal cancer have been identified in prior laboratory studies. By measuring these predefined biomarkers before and after the study intervention, we can assess how they are affected by the intervention, and gain knowledge about their usefulness in colorectal cancer patients on clinical trial.

This study is a Phase IIa clinical biomarker study, using oral aspirin 325 mg taken daily with an arginine-restricted diet designed to reduce arginine intake by at least 30% during the 12-week study period. The biomarkers will be obtained from patient by performing endoscopy (a procedure used to look at the inside of the bowel, rectum and colon) and biopsy (taking samples of tissue), phlebotomy (drawing blood), and urine collection. Biopsies are done to evaluate changes in tissue content that may relate to early events in colon cancer formation. This was the procedure used to diagnose your condition initially. There will be 24 patients enrolled into this study performed through University of California Irvine Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18-80 years of age with a history of surgically removed colon or rectal cancer, and have received treatment for their disease using drugs (adjuvant chemotherapy)
* Subjects must have colon or rectal cancer with stage I, II, or III disease
* Subjects should not have further treatment with radiation therapy. Subjects having already received adjuvant (i.e., post-operative) radiation therapy to the colon or rectum will be excluded. However, subjects receiving radiation therapy prior to surgery for rectal cancer are eligible for enrollment.
* Subject's tumor must have been completely removed within the past 12 months, with first surveillance colonoscopy anticipated 12 weeks after study treatment start date (i.e. one-year after surgical removal).
* Subjects must be in good physical status
* If subjects are premenopausal and perimenopausal women, they must be using adequate birth control methods.
* Subjects must have no history of another invasive cancer within 5 years
* Subjects must have no further chemotherapy anticipated.
* Subjects don't have special dietary requirements or additives. Subjects must not be consuming a diet that would preclude taking the study medication.
* Subjects must have no concomitant use of calcium supplements (> 520mg/day).
* Subjects must have no history of abnormal wound healing or repair, or conditions that predispose to the same.
* Subjects don't have personal history of colon resection of or inflammatory bowel disease.
* Subjects must give informed consent via consent form approved by the local Human Subjects Committee (Institutional Review Board).
* If subjects are taking aspirin 81mg by mouth daily they will be eligible
* Subjects must have no history of allergies or adverse reactions to aspirin.
* Subjects don't have documented history of gastric/duodenal ulcer within the last 12 months.

Exclusion Criteria:

* Subjects already received radiation therapy to the colon or rectum.
* Subjects adhering to vegetarian diets.
* Subjects are pregnant or lactating women.
* Subjects are breastfeeding
* Subjects are already taking aspirin 325mg by mouth daily.
* Subjects are taking combination medication with more than 81mg aspirin.
* Subjects are currently being treated for gastric/duodenal ulcer or experiencing symptoms at study entry.
* Subjects have a history of any medical condition that would place them at risk as a result of a blood donation, they will be excluded from the study.
* Subjects are taking blood-thinning drugs as warfarin (Coumadin)
* Subjects are allergic to fenoprofen, ibuprofen, indomethacin, ketoprofen, meclofenamate sodium, naproxen, sulindac, tolmetin, or an orange food coloring known as tartrazine.
* Subjects have liver damage or severe kidney failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09-24 (Actual); Primary Completion 2013-11-26 (Actual); Study Completion 2013-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Zell, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zell JA, Taylor TH, Albers CG, Carmichael JC, McLaren CE, Wenzel L, Stamos MJ. Phase IIa Clinical Biomarker Trial of Dietary Arginine Restriction and Aspirin in Colorectal Cancer Patients. Cancers (Basel). 2023 Mar 31;15(7):2103. doi: 10.3390/cancers15072103. PMID 37046763

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 325 mg Aspirin
Started | 24
Completed | 20
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | 325 mg Aspirin
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 58 [51.7 to 62.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Rectal Tissue Putrescine Reduction
Description: To demonstrate a > 50% decrease in rectal tissue putrescine levels from baseline in study subjects, as a measure of polyamine reduction in the target tissue of colorectal cancer patients.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 325 mg Aspirin
Number analyzed (Participants) | 20
Participants | 17

2. Secondary Outcome: Safety/Toxicity
Description: To determine the number and proportion of patients with any grade 1 or greater side effect, using Common Terminology for Adverse Events v4.0 (CTCAE)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 325 mg Aspirin
Number analyzed (Participants) | 20
Participants | 6

ADVERSE EVENTS:
Arm/Group | 325 mg Aspirin
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 325 mg Aspirin (N=20)
Diarrhea (General disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Neuropathy (General disorders) | 1 (1)
Myalgia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes